CLINICAL TRIAL: NCT04057820
Title: Eating, Sleeping, Consoling for Neonatal Withdrawal (ESC-NOW): a Function-Based Assessment and Management Approach
Acronym: (ESC-NOW)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advancing Clinical Trials in Neonatal Opioid Withdrawal (ACT NOW) Program (Network)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: ACTNOW-01; 3U2COD023375-06S1 (NIH)
Record Dates: First submitted 2019-08-09; First posted 2019-08-15 (Actual); Results first posted 2023-10-04 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Neonatal Opiate Withdrawal Syndrome
Keywords: NOWS
MeSH Terms: interventions — Eating; Sleep

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized controlled trial with transition period.All sites start with usual care and are transitioned to using the ESC tool
Who Masked: Outcomes Assessor
Masking Description: The protocol study team will assure blinding of the electronically performed follow-up questionnaires through the use of a centralized computer scoring system. However, it will not be possible to blind responses to questionnaires that are performed with the assistance of research personnel at the participating sites. The protocol study team will note the method of questionnaire completion and will evaluate for bias in this context.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care, Finnegan Neonatal Abstinence Scoring Tool (Active Comparator): Usual institutional care for infants with NOWS with the Finnegan Neonatal Abstinence Scoring Tool (FNAST)
  Interventions: Other: Finnegan Neonatal Abstinence Scoring Tool
- Eat, Sleep, Console care tool (Active Comparator): New treatment implemented at the site for infants with NOWS using the Eat, Sleep, Console (ESC) care tool
  Interventions: Other: Eat, Sleep, Console (ESC) care tool

INTERVENTIONS:
Other: Finnegan Neonatal Abstinence Scoring Tool — The FNAST is a scoring system used in neonatal units to initiate and guide therapy in infants of opiate-dependent mothers.
  Other Names: FNAST
  Arms: Usual care, Finnegan Neonatal Abstinence Scoring Tool
Other: Eat, Sleep, Console (ESC) care tool — The ESC care approach emphasizes parental involvement, simplifies the assessment of infants with NOWS and focuses interventions on non-pharmacologic therapies.
  Other Names: ESC
  Arms: Eat, Sleep, Console care tool

SUMMARY:
The overall objective is to determine if the ESC care approach will reduce the time until infants being managed for NOWS are medically ready for discharge.

DETAILED DESCRIPTION:
This study will randomize institutions in blocks to transition from usual institutional care for infants with NOWS to the ESC care approach at a randomly allocated transition period (from usual care to the ESC care approach).

During the initial birth hospitalization, the clinical site research team will collect data under waiver of consent for infants who meet eligibility criteria.

The site research team will obtain informed consent from the legal guardian(s) to obtain long-term outcomes for eligible infants and caregivers. Clinical site research team members may obtain this consent at any point during the hospital stay for infants who meet the trial's inclusion criteria. This data will allow the protocol study team to short- and long-term outcomes for infants managed with the ESC care approach compared to usual institutional care.

ELIGIBILITY:
Inclusion Criteria:

* 1. The infant is being managed for NOWS at an eligible site (i.e., receiving non-pharmacologic care, assessments for withdrawal severity, +/- pharmacologic care) 2. The infant is ≥ 36 weeks gestation 3. The infant satisfies at least 1 of the following criteria:

  1. Maternal history of prenatal opioid use
  2. Maternal toxicology screen positive for opioids during the second and/or third trimester of pregnancy
  3. Infant toxicology screen positive for opioids during the initial hospital stay

Exclusion Criteria:

* 1. Infant has major birth defect(s) 2. Infant has neonatal encephalopathy (inclusive of hypoxic ischemic encephalopathy), a metabolic disorder, stroke, intracranial hemorrhage, or meningitis diagnosed by 60 hours of life 3. Infant was receiving respiratory support (any positive pressure or oxygen therapy) unrelated to pharmacologic treatment for NOWS at 60 hours of life 4. Infant was receiving antimicrobial(s) at 60 hours of life 5. Infant has received any major surgical intervention in the first 60 hours of life 6. Postnatal opioid exposure other than for treatment of NOWS in the first 60 hours of life 7. Outborn infants transferred at >60 hours of life or treated with opioids for NOWS at the transferring hospital

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1305 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2024-09-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Chistiana Care Health Systems, Newark, Delaware
  - Tampa General Hospital, Tampa, Florida
  - Kapiolani Hospital, Honolulu, Hawaii
  - Kansas University Medical Center, Kansas City, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - St. Elizabeth Healthcare/CCHMC, Edgewood, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, Metairie, Louisiana
  - Winchester Hospital, Winchester, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of New Mexico, Albuquerque, New Mexico
  - University of Buffalo, Buffalo, New York
  - University of Rochester, Rochester, New York
  - Duke Hospital, Durham, North Carolina
  - Good Samaritan Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Sanford Health, Sioux Falls, South Dakota
  - University of Utah Medical Center, Salt Lake City, Utah

REFERENCES:
- [Derived] Beauman SGS, Hu Z, Rice W, Devlin L, Merhar SL, Fung CM, Brown J, Osman A, Pahl A, Ramsey KW, Whalen B, MacMillan KDL, Ounpraseuth ST, Das A, Crawford MM, Trochinski L, Greenberg RG, Smith PB, Young LW, Maxwell JR; Eunice Kennedy Shriver NICHD Neonatal Research Network and the NIH ECHO Program IDeA States Pediatrics Clinical Trials Network. Antenatal Exposure to Medication for Opioid Use Disorder and Infant Outcomes in the Eat, Sleep, Console for Neonatal Opioid Withdrawal Randomized Controlled Trial. J Pediatr. 2025 Oct 17;289:114859. doi: 10.1016/j.jpeds.2025.114859. Online ahead of print. PMID 41110632
- [Derived] Merhar SL, Hu Z, Devlin LA, Ounpraseuth ST, Simon AE, Smith PB, Walsh MC, Lee JY, Das A, Higgins RD, Crawford MM, Rice W, Paul DA, Maxwell JR, Telang SD, Fung CM, Wright T, Reynolds AM, Hahn D, Ross J, McAllister JM, Crowley M, Shaikh SK, Christ L, Brown J, Riccio J, Wong Ramsey K, Braswell EF, Tucker L, McAlmon K, Dummula K, Weiner J, White JR, Howell MP, Newman S, Snowden JN, Young LW; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network National Institutes of Health Environmental Influences on Child Health Outcomes Program Institutional Development Award States Pediatric Clinical Tri; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network National Institutes of Health Environmental Influences on Child Health Outcomes Program Institutional Development Award States Pediatric Clinical Trials Network. Infant Feeding and Weight Trajectories in the Eat, Sleep, Console Trial: A Secondary Analysis of a Randomized Clinical Trial. JAMA Pediatr. 2024 Oct 1;178(10):976-984. doi: 10.1001/jamapediatrics.2024.2578. PMID 39133505
- [Derived] Devlin LA, Hu Z, Merhar SL, Ounpraseuth ST, Simon AE, Lee JY, Das A, Crawford MM, Greenberg RG, Smith PB, Higgins RD, Walsh MC, Rice W, Paul DA, Maxwell JR, Fung CM, Wright T, Ross J, McAllister JM, Crowley M, Shaikh SK, Christ L, Brown J, Riccio J, Wong Ramsey K, Braswell EF, Tucker L, McAlmon K, Dummula K, Weiner J, White JR, Newman S, Snowden JN, Young LW; Eunice Kennedy Shriver NICHD Neonatal Research Network and NIH Environmental Influences on Child Health Outcomes (ECHO) Program Institutional Development Award States Pediatric Clinical Trials Network. Influence of Eat, Sleep, and Console on Infants Pharmacologically Treated for Opioid Withdrawal: A Post Hoc Subgroup Analysis of the ESC-NOW Randomized Clinical Trial. JAMA Pediatr. 2024 Jun 1;178(6):525-532. doi: 10.1001/jamapediatrics.2024.0544. PMID 38619854
- [Derived] Young LW, Ounpraseuth ST, Merhar SL, Hu Z, Simon AE, Bremer AA, Lee JY, Das A, Crawford MM, Greenberg RG, Smith PB, Poindexter BB, Higgins RD, Walsh MC, Rice W, Paul DA, Maxwell JR, Telang S, Fung CM, Wright T, Reynolds AM, Hahn DW, Ross J, McAllister JM, Crowley M, Shaikh SK, Puopolo KM, Christ L, Brown J, Riccio J, Wong Ramsey K, Akshatha, Braswell EF, Tucker L, McAlmon KR, Dummula K, Weiner J, White JR, Howell MP, Newman S, Snowden JN, Devlin LA; ACT NOW Collaborative. Eat, Sleep, Console Approach or Usual Care for Neonatal Opioid Withdrawal. N Engl J Med. 2023 Jun 22;388(25):2326-2337. doi: 10.1056/NEJMoa2214470. Epub 2023 Apr 30. PMID 37125831

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The in-hospital and initial follow-up portions of the trial were conducted with a waiver of informed consent, as approved by central institutional review board.
Pre-assignment Details: The in-hospital portion of the study was performed under waiver of informed consent. Only the newborn babies are considered enrolled participants. The number of participants to start a Period may not equal the number who completed a previous Period because at each subsequent Period a new cohort of newborn babies are enrolled at the respective sites. During the transition period for a given block, sites within the block are not enrolling participants.
Units Other Than Participants: Sites
Groups:
- Block 1: Usual Care, Finnegan Neonatal Abstinence Scoring Tool: Usual institutional care for infants with NOWS with the Finnegan Neonatal Abstinence Scoring Tool (FNAST)
  Finnegan Neonatal Abstinence Scoring Tool: The FNAST is a scoring system used in neonatal units to initiate and guide therapy in infants of opiate-dependent mothers.
  Block 1 contained four sites.
- Block 1: Eat, Sleep, Console Care Tool: New treatment implemented at the site for infants with NOWS using the Eat, Sleep, Console (ESC) care tool
  Eat, Sleep, Console (ESC) care tool: The ESC care approach emphasizes parental involvement, simplifies the assessment of infants with NOWS and focuses interventions on non-pharmacologic therapies.
  Block 1 had four sites.
- Block 2: Usual Care, Finnegan Neonatal Abstinence Scoring Tool: Usual institutional care for infants with NOWS with the Finnegan Neonatal Abstinence Scoring Tool (FNAST)
  Finnegan Neonatal Abstinence Scoring Tool: The FNAST is a scoring system used in neonatal units to initiate and guide therapy in infants of opiate-dependent mothers.
  Block 2 contained two sites.
- Block 2: Eat, Sleep, Console Care Tool: New treatment implemented at the site for infants with NOWS using the Eat, Sleep, Console (ESC) care tool
  Eat, Sleep, Console (ESC) care tool: The ESC care approach emphasizes parental involvement, simplifies the assessment of infants with NOWS and focuses interventions on non-pharmacologic therapies.
  Block 2 had two sites.
- Block 3: Usual Care, Finnegan Neonatal Abstinence Scoring Tool: Usual institutional care for infants with NOWS with the Finnegan Neonatal Abstinence Scoring Tool (FNAST)
  Finnegan Neonatal Abstinence Scoring Tool: The FNAST is a scoring system used in neonatal units to initiate and guide therapy in infants of opiate-dependent mothers.
  Block 3 contained three sites.
- Block 3: Eat, Sleep, Console Care Tool: New treatment implemented at the site for infants with NOWS using the Eat, Sleep, Console (ESC) care tool
  Eat, Sleep, Console (ESC) care tool: The ESC care approach emphasizes parental involvement, simplifies the assessment of infants with NOWS and focuses interventions on non-pharmacologic therapies.
  Block 3 had three sites.
- Block 4: Usual Care, Finnegan Neonatal Abstinence Scoring Tool: Usual institutional care for infants with NOWS with the Finnegan Neonatal Abstinence Scoring Tool (FNAST)
  Finnegan Neonatal Abstinence Scoring Tool: The FNAST is a scoring system used in neonatal units to initiate and guide therapy in infants of opiate-dependent mothers.
  Block 4 contained three sites.
- Block 4: Eat, Sleep, Console Care Tool: New treatment implemented at the site for infants with NOWS using the Eat, Sleep, Console (ESC) care tool
  Eat, Sleep, Console (ESC) care tool: The ESC care approach emphasizes parental involvement, simplifies the assessment of infants with NOWS and focuses interventions on non-pharmacologic therapies.
  Block 4 had threesites.
- Block 5: Usual Care, Finnegan Neonatal Abstinence Scoring Tool: Usual institutional care for infants with NOWS with the Finnegan Neonatal Abstinence Scoring Tool (FNAST)
  Finnegan Neonatal Abstinence Scoring Tool: The FNAST is a scoring system used in neonatal units to initiate and guide therapy in infants of opiate-dependent mothers.
  Block 5 contained four sites.
- Block 5: Eat, Sleep, Console Care Tool: New treatment implemented at the site for infants with NOWS using the Eat, Sleep, Console (ESC) care tool
  Eat, Sleep, Console (ESC) care tool: The ESC care approach emphasizes parental involvement, simplifies the assessment of infants with NOWS and focuses interventions on non-pharmacologic therapies.
  Block 5 had four sites.
- Block 6: Usual Care, Finnegan Neonatal Abstinence Scoring Tool: Usual institutional care for infants with NOWS with the Finnegan Neonatal Abstinence Scoring Tool (FNAST)
  Finnegan Neonatal Abstinence Scoring Tool: The FNAST is a scoring system used in neonatal units to initiate and guide therapy in infants of opiate-dependent mothers.
  Block 6 contained four sites.
- Block 6: Eat, Sleep, Console Care Tool: New treatment implemented at the site for infants with NOWS using the Eat, Sleep, Console (ESC) care tool
  Eat, Sleep, Console (ESC) care tool: The ESC care approach emphasizes parental involvement, simplifies the assessment of infants with NOWS and focuses interventions on non-pharmacologic therapies.
  Block 6 had four sites.
- Block 7: Usual Care, Finnegan Neonatal Abstinence Scoring Tool: Usual institutional care for infants with NOWS with the Finnegan Neonatal Abstinence Scoring Tool (FNAST)
  Finnegan Neonatal Abstinence Scoring Tool: The FNAST is a scoring system used in neonatal units to initiate and guide therapy in infants of opiate-dependent mothers.
  Block 7 contained threesites.
- Block 7: Eat, Sleep, Console Care Tool: New treatment implemented at the site for infants with NOWS using the Eat, Sleep, Console (ESC) care tool
  Eat, Sleep, Console (ESC) care tool: The ESC care approach emphasizes parental involvement, simplifies the assessment of infants with NOWS and focuses interventions on non-pharmacologic therapies.
  Block 7 had three sites.
- Block 8: Usual Care, Finnegan Neonatal Abstinence Scoring Tool: Usual institutional care for infants with NOWS with the Finnegan Neonatal Abstinence Scoring Tool (FNAST)
  Finnegan Neonatal Abstinence Scoring Tool: The FNAST is a scoring system used in neonatal units to initiate and guide therapy in infants of opiate-dependent mothers.
  Block 8 contained threesites.
- Block 8: Eat, Sleep, Console Care Tool: New treatment implemented at the site for infants with NOWS using the Eat, Sleep, Console (ESC) care tool
  Eat, Sleep, Console (ESC) care tool: The ESC care approach emphasizes parental involvement, simplifies the assessment of infants with NOWS and focuses interventions on non-pharmacologic therapies.
  Block 8 had three sites.
Period: Period 1
Arm/Group | Block 1: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 1: Eat, Sleep, Console Care Tool | Block 2: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 2: Eat, Sleep, Console Care Tool | Block 3: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 3: Eat, Sleep, Console Care Tool | Block 4: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 4: Eat, Sleep, Console Care Tool | Block 5: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 5: Eat, Sleep, Console Care Tool | Block 6: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 6: Eat, Sleep, Console Care Tool | Block 7: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 7: Eat, Sleep, Console Care Tool | Block 8: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 8: Eat, Sleep, Console Care Tool
Started | 27; 4 Sites | 0; 0 Sites | 8; 2 Sites | 0; 0 Sites | 23; 3 Sites | 0; 0 Sites | 23; 3 Sites | 0; 0 Sites | 41; 4 Sites | 0; 0 Sites | 27; 4 Sites | 0; 0 Sites | 16; 3 Sites | 0; 0 Sites | 20; 3 Sites | 0; 0 Sites
Completed | 27; 4 Sites | 0; 0 Sites | 8; 2 Sites | 0; 0 Sites | 23; 3 Sites | 0; 0 Sites | 23; 3 Sites | 0; 0 Sites | 41; 4 Sites | 0; 0 Sites | 27; 4 Sites | 0; 0 Sites | 16; 3 Sites | 0; 0 Sites | 20; 3 Sites | 0; 0 Sites
Not Completed | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites
Period: Period 2
Arm/Group | Block 1: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 1: Eat, Sleep, Console Care Tool | Block 2: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 2: Eat, Sleep, Console Care Tool | Block 3: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 3: Eat, Sleep, Console Care Tool | Block 4: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 4: Eat, Sleep, Console Care Tool | Block 5: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 5: Eat, Sleep, Console Care Tool | Block 6: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 6: Eat, Sleep, Console Care Tool | Block 7: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 7: Eat, Sleep, Console Care Tool | Block 8: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 8: Eat, Sleep, Console Care Tool
Started | 0; 0 Sites (Block 1 with 4 sites transitioned from Usual Care to ESC during Period 2; therefore no infants were being enrolled and the total number of sites enrolling infants was 22. For this stepped wedge study design, a new cohort of infants is enrolled during each period except the transition period. Therefore, the number of infants to start a period is unlikely to equal the number of infants who completed the previous period.) | 0; 0 Sites | 5; 2 Sites (For this stepped wedge study design, a new cohort of infants is enrolled during each period except the transition period. Therefore, the number of infants to start a period is unlikely to equal the number of infants who completed the previous period.) | 0; 0 Sites | 11; 3 Sites | 0; 0 Sites | 12; 3 Sites | 0; 0 Sites | 47; 4 Sites | 0; 0 Sites | 17; 4 Sites | 0; 0 Sites | 10; 3 Sites | 0; 0 Sites | 18; 3 Sites | 0; 0 Sites
Completed | 0; 0 Sites | 0; 0 Sites | 5; 2 Sites | 0; 0 Sites | 11; 3 Sites | 0; 0 Sites | 12; 3 Sites | 0; 0 Sites | 47; 4 Sites | 0; 0 Sites | 17; 4 Sites | 0; 0 Sites | 10; 3 Sites | 0; 0 Sites | 18; 3 Sites | 0; 0 Sites
Not Completed | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites
Period: Period 3
Arm/Group | Block 1: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 1: Eat, Sleep, Console Care Tool | Block 2: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 2: Eat, Sleep, Console Care Tool | Block 3: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 3: Eat, Sleep, Console Care Tool | Block 4: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 4: Eat, Sleep, Console Care Tool | Block 5: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 5: Eat, Sleep, Console Care Tool | Block 6: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 6: Eat, Sleep, Console Care Tool | Block 7: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 7: Eat, Sleep, Console Care Tool | Block 8: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 8: Eat, Sleep, Console Care Tool
Started | 0; 0 Sites | 25; 4 Sites (For this stepped wedge study design, a new cohort of infants is enrolled during each period except the transition period. Therefore, the number of infants to start a period is unlikely to equal the number of infants who completed the previous period.) | 0; 0 Sites (Block 2 with 2 sites transitioned from Usual Care to ESC during Period 3; therefore no infants were being enrolled and the total number of sites enrolling infants was 24..) | 0; 0 Sites | 7; 3 Sites | 0; 0 Sites | 19; 3 Sites | 0; 0 Sites | 32; 4 Sites | 0; 0 Sites | 15; 4 Sites | 0; 0 Sites | 22; 3 Sites | 0; 0 Sites | 24; 3 Sites | 0; 0 Sites
Completed | 0; 0 Sites | 25; 4 Sites | 0; 0 Sites | 0; 0 Sites | 7; 3 Sites | 0; 0 Sites | 19; 3 Sites | 0; 0 Sites | 32; 4 Sites | 0; 0 Sites | 15; 4 Sites | 0; 0 Sites | 22; 3 Sites | 0; 0 Sites | 24; 3 Sites | 0; 0 Sites
Not Completed | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites
Period: Period 4
Arm/Group | Block 1: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 1: Eat, Sleep, Console Care Tool | Block 2: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 2: Eat, Sleep, Console Care Tool | Block 3: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 3: Eat, Sleep, Console Care Tool | Block 4: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 4: Eat, Sleep, Console Care Tool | Block 5: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 5: Eat, Sleep, Console Care Tool | Block 6: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 6: Eat, Sleep, Console Care Tool | Block 7: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 7: Eat, Sleep, Console Care Tool | Block 8: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 8: Eat, Sleep, Console Care Tool
Started | 0; 0 Sites | 22; 4 Sites (For this stepped wedge study design, a new cohort of infants is enrolled during each period except the transition period. Therefore, the number of infants to start a period is unlikely to equal the number of infants who completed the previous period.) | 0; 0 Sites | 8; 2 Sites | 0; 0 Sites (Block 3 with 3 transitioned from Usual Care to ESC during Period 4; therefore no infants were being enrolled and the total number of sites enrolling infant was 23.) | 0; 0 Sites | 16; 3 Sites | 0; 0 Sites | 33; 4 Sites | 0; 0 Sites | 19; 4 Sites | 0; 0 Sites | 19; 3 Sites | 0; 0 Sites | 22; 3 Sites | 0; 0 Sites
Completed | 0; 0 Sites | 22; 4 Sites | 0; 0 Sites | 8; 2 Sites | 0; 0 Sites | 0; 0 Sites | 16; 3 Sites | 0; 0 Sites | 33; 4 Sites | 0; 0 Sites | 19; 4 Sites | 0; 0 Sites | 19; 3 Sites | 0; 0 Sites | 22; 3 Sites | 0; 0 Sites
Not Completed | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites
Period: Period 5
Arm/Group | Block 1: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 1: Eat, Sleep, Console Care Tool | Block 2: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 2: Eat, Sleep, Console Care Tool | Block 3: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 3: Eat, Sleep, Console Care Tool | Block 4: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 4: Eat, Sleep, Console Care Tool | Block 5: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 5: Eat, Sleep, Console Care Tool | Block 6: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 6: Eat, Sleep, Console Care Tool | Block 7: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 7: Eat, Sleep, Console Care Tool | Block 8: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 8: Eat, Sleep, Console Care Tool
Started | 0; 0 Sites | 25; 4 Sites (For this stepped wedge study design, a new cohort of infants is enrolled during each period except the transition period. Therefore, the number of infants to start a period is unlikely to equal the number of infants who completed the previous period.) | 0; 0 Sites | 8; 2 Sites | 0; 0 Sites | 12; 3 Sites | 0; 0 Sites (Block 4 with 3 sites transitioned from Usual Care to ESC during Period 5; therefore no infants were being enrolled and the total number of sites enrolling infants was 23.) | 0; 0 Sites | 16; 4 Sites | 0; 0 Sites | 19; 4 Sites | 0; 0 Sites | 16; 3 Sites | 0; 0 Sites | 17; 3 Sites | 0; 0 Sites
Completed | 0; 0 Sites | 25; 4 Sites | 0; 0 Sites | 8; 2 Sites | 0; 0 Sites | 12; 3 Sites | 0; 0 Sites | 0; 0 Sites | 16; 4 Sites | 0; 0 Sites | 19; 4 Sites | 0; 0 Sites | 16; 3 Sites | 0; 0 Sites | 17; 3 Sites | 0; 0 Sites
Not Completed | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites
Period: Period 6
Arm/Group | Block 1: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 1: Eat, Sleep, Console Care Tool | Block 2: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 2: Eat, Sleep, Console Care Tool | Block 3: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 3: Eat, Sleep, Console Care Tool | Block 4: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 4: Eat, Sleep, Console Care Tool | Block 5: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 5: Eat, Sleep, Console Care Tool | Block 6: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 6: Eat, Sleep, Console Care Tool | Block 7: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 7: Eat, Sleep, Console Care Tool | Block 8: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 8: Eat, Sleep, Console Care Tool
Started | 0; 0 Sites | 24; 4 Sites (For this stepped wedge study design, a new cohort of infants is enrolled during each period except the transition period. Therefore, the number of infants to start a period is unlikely to equal the number of infants who completed the previous period.) | 0; 0 Sites | 5; 2 Sites | 0; 0 Sites | 14; 3 Sites | 0; 0 Sites | 15; 3 Sites | 0; 0 Sites (Block 5 with 4 sites transitioned from Usual Care to ESC during Period 6; therefore no infants were being enrolled and the total number of sites enrolling infants was 22.) | 0; 0 Sites | 13; 4 Sites | 0; 0 Sites | 17; 3 Sites | 0; 0 Sites | 18; 3 Sites | 0; 0 Sites
Completed | 0; 0 Sites | 24; 4 Sites | 0; 0 Sites | 5; 2 Sites | 0; 0 Sites | 14; 3 Sites | 0; 0 Sites | 15; 3 Sites | 0; 0 Sites | 0; 0 Sites | 13; 4 Sites | 0; 0 Sites | 17; 3 Sites | 0; 0 Sites | 18; 3 Sites | 0; 0 Sites
Not Completed | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites
Period: Period 7
Arm/Group | Block 1: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 1: Eat, Sleep, Console Care Tool | Block 2: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 2: Eat, Sleep, Console Care Tool | Block 3: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 3: Eat, Sleep, Console Care Tool | Block 4: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 4: Eat, Sleep, Console Care Tool | Block 5: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 5: Eat, Sleep, Console Care Tool | Block 6: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 6: Eat, Sleep, Console Care Tool | Block 7: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 7: Eat, Sleep, Console Care Tool | Block 8: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 8: Eat, Sleep, Console Care Tool
Started | 0; 0 Sites | 24; 4 Sites | 0; 0 Sites | 9; 2 Sites | 0; 0 Sites | 14; 3 Sites | 0; 0 Sites | 15; 3 Sites | 0; 0 Sites | 34; 4 Sites | 0; 0 Sites (Block 6 with 4 sites transitioned from Usual Care to ESC during Period 7; therefore no infants were being enrolled and the total number of sites enrolling infants was 22.) | 0; 0 Sites | 12; 3 Sites | 0; 0 Sites | 19; 3 Sites | 0; 0 Sites
Completed | 0; 0 Sites | 24; 4 Sites | 0; 0 Sites | 9; 2 Sites | 0; 0 Sites | 14; 3 Sites | 0; 0 Sites | 15; 3 Sites | 0; 0 Sites | 34; 4 Sites | 0; 0 Sites | 0; 0 Sites | 12; 3 Sites | 0; 0 Sites | 19; 3 Sites | 0; 0 Sites
Not Completed | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites
Period: Period 8
Arm/Group | Block 1: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 1: Eat, Sleep, Console Care Tool | Block 2: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 2: Eat, Sleep, Console Care Tool | Block 3: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 3: Eat, Sleep, Console Care Tool | Block 4: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 4: Eat, Sleep, Console Care Tool | Block 5: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 5: Eat, Sleep, Console Care Tool | Block 6: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 6: Eat, Sleep, Console Care Tool | Block 7: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 7: Eat, Sleep, Console Care Tool | Block 8: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 8: Eat, Sleep, Console Care Tool
Started | 0; 0 Sites | 21; 4 Sites (For this stepped wedge study design, a new cohort of infants is enrolled during each period except the transition period. Therefore, the number of infants to start a period is unlikely to equal the number of infants who completed the previous period.) | 0; 0 Sites | 10; 2 Sites | 0; 0 Sites | 14; 3 Sites | 0; 0 Sites | 18; 3 Sites | 0; 0 Sites | 32; 4 Sites | 0; 0 Sites | 9; 4 Sites | 0; 0 Sites (Block 7 with 3 sites transitioned from Usual Care to ESC during Period 8; therefore no infants were being enrolled and the total number of sites enrolling infants was 23.) | 0; 0 Sites | 22; 3 Sites | 0; 0 Sites
Completed | 0; 0 Sites | 21; 4 Sites | 0; 0 Sites | 10; 2 Sites | 0; 0 Sites | 14; 3 Sites | 0; 0 Sites | 18; 3 Sites | 0; 0 Sites | 32; 4 Sites | 0; 0 Sites | 9; 4 Sites | 0; 0 Sites | 0; 0 Sites | 22; 3 Sites | 0; 0 Sites
Not Completed | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites
Period: Period 9
Arm/Group | Block 1: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 1: Eat, Sleep, Console Care Tool | Block 2: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 2: Eat, Sleep, Console Care Tool | Block 3: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 3: Eat, Sleep, Console Care Tool | Block 4: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 4: Eat, Sleep, Console Care Tool | Block 5: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 5: Eat, Sleep, Console Care Tool | Block 6: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 6: Eat, Sleep, Console Care Tool | Block 7: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 7: Eat, Sleep, Console Care Tool | Block 8: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 8: Eat, Sleep, Console Care Tool
Started | 0; 0 Sites | 18; 4 Sites (For this stepped wedge study design, a new cohort of infants is enrolled during each period except the transition period. Therefore, the number of infants to start a period is unlikely to equal the number of infants who completed the previous period.) | 0; 0 Sites | 3; 2 Sites | 0; 0 Sites | 5; 3 Sites | 0; 0 Sites | 17; 3 Sites | 0; 0 Sites | 28; 4 Sites | 0; 0 Sites | 15; 4 Sites | 0; 0 Sites | 14; 3 Sites | 0; 0 Sites (Block 8 with 3 sites transitioned from Usual Care to ESC during Period 9; therefore no infants were being enrolled and the total number of sites enrolling infants was 23.) | 0; 0 Sites
Completed | 0; 0 Sites | 18; 4 Sites | 0; 0 Sites | 3; 2 Sites | 0; 0 Sites | 5; 3 Sites | 0; 0 Sites | 17; 3 Sites | 0; 0 Sites | 28; 4 Sites | 0; 0 Sites | 15; 4 Sites | 0; 0 Sites | 14; 3 Sites | 0; 0 Sites | 0; 0 Sites
Not Completed | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites
Period: Period 10
Arm/Group | Block 1: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 1: Eat, Sleep, Console Care Tool | Block 2: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 2: Eat, Sleep, Console Care Tool | Block 3: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 3: Eat, Sleep, Console Care Tool | Block 4: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 4: Eat, Sleep, Console Care Tool | Block 5: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 5: Eat, Sleep, Console Care Tool | Block 6: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 6: Eat, Sleep, Console Care Tool | Block 7: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 7: Eat, Sleep, Console Care Tool | Block 8: Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Block 8: Eat, Sleep, Console Care Tool
Started | 0; 0 Sites | 26; 4 Sites (For this stepped wedge study design, a new cohort of infants is enrolled during each period except the transition period. Therefore, the number of infants to start a period is unlikely to equal the number of infants who completed the previous period.) | 0; 0 Sites | 8; 2 Sites | 0; 0 Sites | 17; 3 Sites | 0; 0 Sites | 7; 3 Sites | 0; 0 Sites | 32; 4 Sites | 0; 0 Sites | 17; 4 Sites | 0; 0 Sites | 23; 3 Sites | 0; 0 Sites | 15; 3 Sites
Completed | 0; 0 Sites | 26; 4 Sites | 0; 0 Sites | 8; 2 Sites | 0; 0 Sites | 17; 3 Sites | 0; 0 Sites | 7; 3 Sites | 0; 0 Sites | 32; 4 Sites | 0; 0 Sites | 17; 4 Sites | 0; 0 Sites | 23; 3 Sites | 0; 0 Sites | 15; 3 Sites
Not Completed | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Eat, Sleep, Console Care Tool | Total
Number analyzed (Participants) | 702 | 603 | 1305
Age, Continuous [Mean (Standard Deviation); unit: years] — This information represents maternal age. Population: There were 11 observations with missing maternal age in the Usual Care group while the ESC group had 2 missing maternal age values.
  years
    number analyzed (Participants) | 691 | 601 | 1292
    (all) | 30.4 (4.7) | 31.0 (4.7) | 30.7 (4.7)
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Gestational age at birth
  weeks | 38.6 (1.3) | 38.6 (1.3) | 38.6 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants] — This information represents the infant's sex.
  Participants
    Female | 336 | 314 | 650
    Male | 366 | 289 | 655
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 702 | 603 | 1305
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 107 | 33 | 140
  Not Hispanic or Latino | 576 | 538 | 1114
  Unknown or Not Reported | 19 | 32 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 4 | 16
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 4 | 11 | 15
  Black or African American | 104 | 72 | 176
  White | 555 | 480 | 1035
  More than one race | 1 | 6 | 7
  Unknown or Not Reported | 24 | 27 | 51
Region of Enrollment [Number; unit: participants]
  United States | 702 | 603 | 1305
Marital Status [Count of Participants; unit: Participants]
  Married | 99 | 101 | 200
  Single | 582 | 492 | 1074
  Unknown | 21 | 10 | 31
Gravidity [Median (Inter-Quartile Range); unit: Pregnancies] — Population: There was one observation in the Usual Care group with missing gravidity value.
  Pregnancies
    number analyzed (Participants) | 701 | 603 | 1304
    (all) | 3 [2 to 5] | 4 [2 to 5] | 4 [2 to 5]
Parity [Median (Inter-Quartile Range); unit: Births] — Population: There was one observation in the Usual Care group with missing parity value.
  Births
    number analyzed (Participants) | 701 | 603 | 1304
    (all) | 3 [2 to 4] | 3 [2 to 4] | 3 [2 to 4]
Highest Level of Education [Count of Participants; unit: Participants]
  8th grade or less | 8 | 6 | 14
  9th grade to 12th grade | 69 | 50 | 119
  High school diploma | 125 | 99 | 224
  Partial college or Associate's degree | 69 | 50 | 119
  College degree | 7 | 9 | 16
  Trade or Technical School | 2 | 0 | 2
  Graduate degree | 2 | 3 | 5
  Unknown | 420 | 386 | 806
Mother's Medical Insurance [Number; unit: participants] — Medical insurance is a check "all that applies" question; therefore, the total number may exceed the group sample size.
  participants
    Public Insurance | 633 | 521 | 1154
    Private | 47 | 67 | 114
    Self-pay/uninsured | 18 | 11 | 29
    Other | 0 | 3 | 3
    Unknown | 21 | 8 | 29
Infant weight at birth [Mean (Standard Deviation); unit: g] | 3026.4 (445.4) | 3012.8 (490.4) | 3020.1 (471.8)
Head circumference at birth [Mean (Standard Deviation); unit: cm] — Infant head circumference at birth Population: In the Usual Care group, 10 infants had missing head circumference values while 12 infants had missing observations in the ESC group.
  cm
    number analyzed (Participants) | 692 | 591 | 1283
    (all) | 33.4 (1.9) | 33.5 (1.7) | 33.4 (1.8)
Length at birth [Mean (Standard Deviation); unit: cm] — This represents the infant's length at birth. Population: There were 4 infants in the Usual Care group with missing length at birth while 7 infants in the ESC group had missing observations.
  cm
    number analyzed (Participants) | 698 | 596 | 1294
    (all) | 48.8 (2.6) | 48.8 (2.8) | 48.8 (2.7)
1-minute Apgar scores [Median (Inter-Quartile Range); unit: Score on a scale] — Population: Apgar stands for Appearance, Pulse, Grimace, Activity and Respiration with 5 categories (breathing effort, heart rate, muscle tone, reflexes, skin color) each measured on a scale of 0, 1, 2 (range 0 to 10 with higher scores representing better outcome).
  The 1-minute evaluation is used to determine how well the infant tolerated the birthing process.
  There were 13 infants with missing 1-min Apgar scores in the Usual Care group while 9 infants had missing observations in the ESC group.
  Score on a scale
    number analyzed (Participants) | 689 | 594 | 1283
    (all) | 8 [8 to 8] | 8 [8 to 8] | 8 [8 to 8]
5-minute Apgar scores [Median (Inter-Quartile Range); unit: Score on a scale] — Population: Apgar stands for Appearance, Pulse, Grimace, Activity and Respiration with 5 categories (breathing effort, heart rate, muscle tone, reflexes, skin color) each measured on a scale of 0, 1, 2 (range 0 to 10 with higher scores representing better outcome).
  The 5-minute score measures how well the infant is doing outside the mother's womb.
  There were 14 infants with missing 5-min Apgar scores in the Usual Care group while 7 infants had missing observations in the ESC group.
  Score on a scale
    number analyzed (Participants) | 688 | 596 | 1284
    (all) | 9 [9 to 9] | 9 [9 to 9] | 9 [9 to 9]
10-minute Apgar scores [Median (Inter-Quartile Range); unit: Score on a scale] — Population: Apgar stands for Appearance, Pulse, Grimace, Activity and Respiration with 5 categories (breathing effort, heart rate, muscle tone, reflexes, skin color) each measured on a scale of 0, 1, 2 (range 0 to 10 with higher scores representing better outcome).
  The Usual Care group had 668 infants with missing 10-min Apgar scores while ESC had 574 missing 10-min Apgar scores.
  Score on a scale
    number analyzed (Participants) | 34 | 29 | 63
    (all) | 8 [8 to 9] | 9 [8 to 9] | 8 [8 to 9]

OUTCOME MEASURES:

1. Primary Outcome: Time From Birth Until Medically Ready for Discharge
Description: The number of days from birth until the infant is determined to be medically ready for discharge per protocol. The criteria for medical readiness were prospectively defined as an age of at least 96 hours, a period of at least 48 hours without receipt of an opioid, at least 24 hours with no respiratory support and with 100% oral feeding, and at least 24 hours from initiation of maximum caloric density.
Time Frame: from date of birth until hospital discharge or 1 year whichever comes first
Population: The primary analysis population only included those infants that met the definition of medically ready for discharge.
Measure: Least Squares Mean (95% Confidence Interval); unit: days
Arm/Group | Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Eat, Sleep, Console Care Tool
Number analyzed (Participants) | 440 | 397
days | 14.9 [13.1 to 16.7] | 8.2 [7.2 to 9.2]
Statistical Analysis 1: Comparison: Usual Care, Finnegan Neonatal Abstinence Scoring Tool vs Eat, Sleep, Console Care Tool; Test type: Superiority; p < 0.0001, Mixed Models Analysis; The model adjusted for study design (i.e., fixed time effect and random site effect) and randomization scheme stratification indicator; Incidence rate ratio (IRR) = 0.55, 95% CI 2-sided [0.46 to 0.65]

2. Secondary Outcome: Did Infant Receive Opioid Replacement Therapy (Yes/no)
Description: Review of hospital records to determine if infant received opioid replacement therapy prior to hospital discharge
Time Frame: From date of birth until hospital discharge or 1 year whichever comes first
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Eat, Sleep, Console Care Tool
Number analyzed (Participants) | 702 | 603
Participants | 328 | 145
Statistical Analysis 1: Comparison: Usual Care, Finnegan Neonatal Abstinence Scoring Tool vs Eat, Sleep, Console Care Tool; Test type: Superiority; p < 0.0001, Mixed-effect Poisson w/ robust err var; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.38, 95% CI 2-sided [0.30 to 0.47]

3. Secondary Outcome: Total Dose of Opioid Replacement Therapy Infant Received
Description: If infant received opioid replacement therapy, the units received (mg/kg).
Time Frame: From date of birth until hospital discharge or 1 year whichever comes first
Population: The analysis population for this outcome include only infants who received opioid treatment.
Measure: Mean (95% Confidence Interval); unit: mg/kg
Arm/Group | Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Eat, Sleep, Console Care Tool
Number analyzed (Participants) | 324 | 144
mg/kg | 7.5 [5.0 to 10.1] | 5.3 [3.2 to 7.4]
Statistical Analysis 1: Comparison: Usual Care, Finnegan Neonatal Abstinence Scoring Tool vs Eat, Sleep, Console Care Tool; Test type: Superiority; Mean Difference (Final Values) = 2.3, 95% CI 2-sided [-0.4 to 4.9]

4. Secondary Outcome: Time Until Initiation of Opioid Replacement
Description: If infant received opioid replacement therapy, the timing of the initiation of therapy
Time Frame: From date of birth until hospital discharge or 1 year whichever comes first
Population: The analysis population for this outcome include only infants who received opioid treatment.
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Eat, Sleep, Console Care Tool
Number analyzed (Participants) | 324 | 144
hours | 53.0 [48.7 to 57.3] | 76 [63.0 to 89.0]
Statistical Analysis 1: Comparison: Usual Care, Finnegan Neonatal Abstinence Scoring Tool vs Eat, Sleep, Console Care Tool; Test type: Superiority; Mean Difference (Final Values) = 23.0, 95% CI 2-sided [8.1 to 37.9]

5. Secondary Outcome: Receipt of Adjuvant Therapy
Description: To see if the infant had to have any other type of therapy for NOWS (yes/no)
Time Frame: from date of birth until hospital discharge or 1 year whichever comes first
Population: The analysis population for this outcome include only infants who received opioid treatment.
Measure: Number (95% Confidence Interval); unit: percentage who received adjuvant therapy
Arm/Group | Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Eat, Sleep, Console Care Tool
Number analyzed (Participants) | 324 | 144
percentage who received adjuvant therapy | 19.4 [8.5 to 30.4] | 15.7 [5.5 to 25.8]
Statistical Analysis 1: Comparison: Usual Care, Finnegan Neonatal Abstinence Scoring Tool vs Eat, Sleep, Console Care Tool; Test type: Superiority; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.37 to 1.76]

6. Secondary Outcome: Maximum Percent Change in Weight During Initial Birth Hospitalization
Description: Assess percent change in birthweight during hospitalization (i.e., [minimum weight - birth weight] / birth weight)
Time Frame: from date of birth until hospital discharge or 1 year whichever comes first
Measure: Mean (95% Confidence Interval); unit: percentage of change in birth weight
Arm/Group | Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Eat, Sleep, Console Care Tool
Number analyzed (Participants) | 702 | 603
percentage of change in birth weight | 7.6 [7.2 to 8.0] | 8.0 [7.5 to 8.4]
Statistical Analysis 1: Comparison: Usual Care, Finnegan Neonatal Abstinence Scoring Tool vs Eat, Sleep, Console Care Tool; Test type: Superiority; Mixed Models Analysis; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.3 to 1.0]

7. Secondary Outcome: Feeding Type at Discharge (Exclusive Maternal Breast Milk)
Description: Exclusive maternal breast milk feeding at the time of hospital discharge
Time Frame: from date of birth until hospital discharge or 1 year whichever comes first
Measure: Number (95% Confidence Interval); unit: percentage of exclusive breast milk
Arm/Group | Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Eat, Sleep, Console Care Tool
Number analyzed (Participants) | 702 | 603
percentage of exclusive breast milk | 6.3 [2.7 to 9.8] | 12.1 [7.2 to 17.1]
Statistical Analysis 1: Comparison: Usual Care, Finnegan Neonatal Abstinence Scoring Tool vs Eat, Sleep, Console Care Tool; Test type: Superiority; Risk Ratio (RR) = 1.94, 95% CI 2-sided [0.94 to 3.99]

8. Secondary Outcome: Any Direct Breast Feeding at Discharge
Description: Direct breastfeeding within 24 hours of hospital discharge (yes/no)
Time Frame: within 24 hours of hospital discharge
Measure: Number (95% Confidence Interval); unit: percentage of direct breast feeding
Arm/Group | Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Eat, Sleep, Console Care Tool
Number analyzed (Participants) | 702 | 603
percentage of direct breast feeding | 19.5 [15.3 to 23.7] | 32.7 [23.2 to 42.2]
Statistical Analysis 1: Comparison: Usual Care, Finnegan Neonatal Abstinence Scoring Tool vs Eat, Sleep, Console Care Tool; Test type: Superiority; Risk Ratio (RR) = 1.68, 95% CI 2-sided [1.13 to 2.48]

9. Secondary Outcome: Length of Hospital Stay
Description: Time from birth until infants being managed for NOWS are discharged from the hospital
Time Frame: from date of birth until hospital discharge or 1 year whichever comes first
Measure: Least Squares Mean (95% Confidence Interval); unit: days
Arm/Group | Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Eat, Sleep, Console Care Tool
Number analyzed (Participants) | 702 | 603
days | 14.0 [12.7 to 15.3] | 7.8 [7.1 to 8.5]
Statistical Analysis 1: Comparison: Usual Care, Finnegan Neonatal Abstinence Scoring Tool vs Eat, Sleep, Console Care Tool; Test type: Superiority; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Incidence ratio ratio (IRR) = 0.56, 95% CI 2-sided [0.49 to 0.64]

10. Secondary Outcome: Inpatient Composite Safety Outcome Which Includes Seizures, Accidental Trauma, Respiratory Insufficiency Due to Opioid Therapy (Present/Absent)
Description: composite of the following: seizures, accidental trauma, respiratory insufficiency due to opioid therapy
Time Frame: from date of birth until hospital discharge or 1 year whichever comes first
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Eat, Sleep, Console Care Tool
Number analyzed (Participants) | 702 | 603
Participants | 1 | 2

11. Secondary Outcome: Composite of the Following: Acute/Urgent Care and/or Emergency Room Visits, Hospital Readmissions
Description: Outpatient composite safety outcome which includes acute/urgent care and/or emergency room visits, hospital readmissions at 3 months (present/absent)
Time Frame: at 3 months of age
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Eat, Sleep, Console Care Tool
Number analyzed (Participants) | 702 | 603
Participants | 113 | 86
Statistical Analysis 1: Comparison: Usual Care, Finnegan Neonatal Abstinence Scoring Tool vs Eat, Sleep, Console Care Tool; Test type: Superiority; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.71 to 1.47]

12. Secondary Outcome: Critical Safety Outcome
Description: any non-accidental trauma and death (yes/no)
Time Frame: at 3 months of age.
Measure: Number; unit: number of non-accidental trauma/death
Arm/Group | Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Eat, Sleep, Console Care Tool
Number analyzed (Participants) | 702 | 603
number of non-accidental trauma/death | 5 | 1

ADVERSE EVENTS:
Time Frame: 3-months post-hospital discharge
Arm/Group | Usual Care, Finnegan Neonatal Abstinence Scoring Tool | Eat, Sleep, Console Care Tool
All-Cause Mortality (participants affected / at risk) | 4/702 | 0/603
Serious Adverse Events (participants affected / at risk) | 4/702 | 12/603
Other Adverse Events (participants affected / at risk) | 8/702 | 18/603
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care, Finnegan Neonatal Abstinence Scoring Tool (N=702) | Eat, Sleep, Console Care Tool (N=603)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) — SAE during main study in-hospital prior to discharge.
Severe Weight Loss (Metabolism and nutrition disorders) | 0 (0) | 2 (2) — SAE during main study in-hospital prior to discharge.
Accidental trauma (infant dropped) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — SAE during main study in-hospital prior to discharge.
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — SAE reported after discharge from hospital.
Accidental Drug Ingestion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — SAE reported after discharge from hospital.
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 1 (1) — SAE reported after discharge from hospital.
Poor weight gain (Metabolism and nutrition disorders) | 1 (1) | 1 (1) — SAE reported after discharge from hospital.
Abnormal echocardiogram (Cardiac disorders) | 0 (0) | 1 (1) — SAE reported after discharge from hospital.
Acute Covid-19 (Infections and infestations) | 0 (0) | 1 (1) — SAE reported after discharge from hospital.
Tachypnea required readmission to hospital (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — SAE reported after discharge from hospital.
Ventricular Septal Defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) — SAE reported after discharge from hospital.
Viral Meningitis (Infections and infestations) | 0 (0) | 1 (1) — SAE reported after discharge from hospital.
Vomiting R11.10 (Gastrointestinal disorders) | 0 (0) | 1 (1) — SAE reported after discharge from hospital.
Observation and evaluation of newborn sepsis (Infections and infestations) | 0 (0) | 1 (1) — SAE reported after discharge from hospital.
Severe Weight Loss (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — SAE reported after discharge from hospital.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care, Finnegan Neonatal Abstinence Scoring Tool (N=702) | Eat, Sleep, Console Care Tool (N=603)
Severe Weight Loss (Metabolism and nutrition disorders) | 5 (5) | 12 (12) — AE during main study in-hospital prior to discharge.
Accidental trauma (infant dropped) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — AE during main study in-hospital prior to discharge.
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) — AE during main study in-hospital prior to discharge.
CMV (Infections and infestations) | 0 (0) | 2 (2) — AE during main study in-hospital prior to discharge.
Fall, caught before hitting floor (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — AE during main study in-hospital prior to discharge.
Diaper Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — AE during main study after hospital discharge.
Non-accidental trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — AE during main study after hospital discharge.
PCP suspected resp. distress, not confirmed by ED (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — AE during main study after hospital discharge.
Frequent emesis (Gastrointestinal disorders) | 0 (0) | 1 (1) — AE during main study after hospital discharge.
Neonatal sleep myoclonus (Nervous system disorders) | 0 (0) | 1 (1) — AE during main study after hospital discharge.
Attention to g-tube (Gastrointestinal disorders) | 0 (0) | 1 (1) — AE during main study after hospital discharge.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (5):
  • Study Protocol and Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT04057820/Prot_SAP_000.pdf
  • Informed Consent Form: General Consent (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/20/NCT04057820/ICF_001.pdf
  • Informed Consent Form: Consent for parent and minor mother (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/20/NCT04057820/ICF_002.pdf
  • Informed Consent Form: Consent for caregiver only (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT04057820/ICF_003.pdf
  • Informed Consent Form: Consent for baby only (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT04057820/ICF_004.pdf